CLINICAL TRIAL: NCT00858494
Title: Homeopathic Cold Medicine for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Standard Homeopathic Company (Industry)
Responsible Party: Principal Investigator, James Taylor, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35537
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Upper Respiratory Tract Infection
Keywords: upper respiratory tract infection; children; homeopathic
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- homeopathic cold remedy (Experimental)
  Interventions: Drug: Hyland's Cold 'n Cough 4 Kids

INTERVENTIONS:
Drug: Hyland's Cold 'n Cough 4 Kids — Liquid homeopathic cold remedy, 5 ml by mouth every 4 hours as needed for relief of cold symptoms for up to 10 days

SUMMARY:
The purpose of this study is to determine if a commercially available homeopathic cold remedy for children is effective in providing relief from cold symptoms in children 2-5 years old. It is postulated that children will have relief of symptoms after receiving a dose of the cold remedy

ELIGIBILITY:
Inclusion Criteria:

* Children 24-59 months old
* Cold/cough symptoms of <7 days duration
* Diagnosed with upper respiratory tract infection by physician or nurse practitioner
* Parent who speaks and reads English

Exclusion Criteria:

* Use of chronic medication other than multivitamins
* History of asthma
* Medication other than acetaminophen or ibuprofen
* Use of homeopathic remedy within preceding 30 days
* Only 1 participant per family

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center-Roosevelt Pediatric Care Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children diagnosed with an upper respiratory tract infection (URI) at a pediatric clinic were recruited for the study from March to September 2009
Pre-assignment Details: one participant who was enrolled had a positive test for streptococcal pharyngitis at the index visit and was prescribed antibiotics. This participant thus became ineligible.
Groups:
- Homeopathic Cold Remedy: Hyland's Cold 'n Cough for Kids, 5 ml by mouth up to 6 times per day as needed for cold symptoms
Period: Overall Study
Arm/Group | Homeopathic Cold Remedy
Started | 49
Completed | 45 (2 participants dropped out before giving study medication. Symptoms resolved without a dose in 2.)
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Homeopathic Cold Remedy
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.5 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Relief of Upper Respiratory Tract Infection (URI) Symptoms (Cough, Runny Nose, Nasal Congestion, Sneezing)1 Hour After Dose of Homeopathic Remedy.
Description: For each dose of study medication, parents indicated which of the symptoms were present (runny nose, cough, nasal congestion, sneezing). Parents rated change in each symptom present one hour after a dose of study medication for up to 6 doses in study logs. Responses were dichotomized as at least some improvement or better (improvement) vs. no improvement or worse. The outcome measure is number of times that improvement in a specific symptom was noted after a dose of the homeopathic remedy. Completed study logs were received from 37 of 49 enrolled participants.
Time Frame: up to 10 days from index visit
Population: Some symptoms were not present at each dose of the homeopathic remedy. Number of doses at which symptom was present: runny nose: 135, nasal congestion: 152, cough: 154, sneezing 81. The outcome is number of times improvement in each symptom was noted.
Measure: Number; unit: doses
Units Other Than Participants: doses
Arm/Group | Homeopathic Cold Remedy
Number analyzed (Participants) | 37
Number analyzed (doses) | 179
doses
  Runny Nose (treated with 135 doses) | 83
  Cough (treated with 154 doses) | 100
  Nasal congestion (treated with 152 doses) | 94
  Sneezing (treated with 81 doses) | 52

2. Secondary Outcome: Parental Report of an Adverse Event After a Dose of Study Medication
Description: After each dose of study medication parents reported the presence of any adverse events
Time Frame: data collected after doses occurring up to 10 days after index visit
Population: Study logs were returned in 37 of 49 enrolled participants. After each dose of study medication, the participant's parent indicated in the study log whether any adverse events were noted.
Measure: Number; unit: doses
Units Other Than Participants: doses
Arm/Group | Homeopathic Cold Remedy
Number analyzed (Participants) | 37
Number analyzed (doses) | 179
doses
  any adverse event | 3
  diarrhea | 2
  excessive gas | 1

ADVERSE EVENTS:
Time Frame: up to 10 days after the index visit
Description: Parents noted any adverse events after each dose of study medication in study logs that were returned to the research staff. Data on any adverse event were based on information in study logs returned in 37 of 49 participants. Parents were instructed to call research team if a serious adverse event occurred; data on all 49 participants presented.
Arm/Group | Homeopathic Cold Remedy
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 2/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Homeopathic Cold Remedy (N=37)
diarrhea (Gastrointestinal disorders) | 1 (2) — Parent noted diarrhea after 2 doses of study medication (occurred in 1 child)
excessive gas (Gastrointestinal disorders) | 1 (1) — parent noted excessive gas after 1 dose of study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less